CLINICAL TRIAL: NCT07225621
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial Comparing Standard of Care Adjuvant Temozolomide With or Without 5-Aminolevulinic Acid (5-ALA) With Concomitant Low Intensity Diffuse Ultrasound (LIDU) Sonodynamic Therapy (SDT) System In Patients With Newly Diagnosed Glioblastoma After Completion of Chemoradiotherapy
Brief Title: Adjuvant Temozolomide ± 5-Aminolevulinic Acid + Low Intensity Diffuse Ultrasound Sonodynamic Therapy System for Newly Diagnosed Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alpheus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV01-201
Record Dates: First submitted 2025-10-30; First posted 2025-11-06 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma; GBM
MeSH Terms: conditions — Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: (experimental arm) (Experimental): * 5-ALA HCl (5-amino-levulenic acid) for oral solution (20 mg/kg) p.o. 6-8 hours prior to LIDU SDT
  * LIDU SDT System (low intensity diffuse ultrasound sonodynamic therapy), for 40 minutes followed by standard of care TMZ
  * SOC TMZ to be started Day 2 (+/-1 day) per the approved PI
  Interventions: Combination Product: 5-ALA HCl + LIDU SDT
- Arm B: (placebo arm) (Placebo Comparator): * Placebo oral solution (matched to 20 mg/kg) p.o. 6-8 hours prior to Sham SDT
  * Sham SDT for 40 mimnutes followed by standard of care TMZ
  * SOC TMZ to be started Day 2 (+/-1 day) per the approved PI
  Interventions: Combination Product: Placebo + Sham SDT

INTERVENTIONS:
Combination Product: 5-ALA HCl + LIDU SDT — standard of care temozolomide + sonosenitizer + sonodynamic therapy
  Arms: Arm A: (experimental arm)
Combination Product: Placebo + Sham SDT — standard of care temozolomide + placebo + sham sonodynamic therapy
  Arms: Arm B: (placebo arm)

SUMMARY:
The purpose of this research is to test an investigational device using ultrasound along with an investigational drug to see if it is useful in treating glioblastoma following standard of care therapy surgery and chemoradiation. This study is evaluating an experimental treatment for glioblastoma that uses an investigational drug (5-ALA) combined with a non-invasive ultrasound device (LIDU) to target tumor cells. Patients meeting the entry requirements to be in the study, will be equally randomly assigned to receive the study device plus the active study drug plus active ultrasound, or to a "sham" procedure where the ultrasound is not being activated and the study drug is a placebo (looks the same but does not contain active drug). Neither the patient or the investigator will know who is in the active group or not. Both groups will continue to receive the standard therapy of oral Temozolomide.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must provide informed consent, stating understanding of the procedures and investigational nature of the study treatment, and willingness to comply with study requirements
2. ≥ 18 and ≤ 80 years of age
3. WHO performance status of ≤ 2 at screening
4. Newly diagnosed Histologically proven glioblastoma (WHO criteria 2021), absence of IDH mutation demonstrated by negative IDH1 R132H staining on Immunohistochemistry.
5. GBM patients that have an absence of disease progression post craniotomy and TMZ/RT. Note: patients must have undergone prior tumor resection to the extent safely feasible (biopsy only are not eligible).
6. Completion of chemoradiation consisting of radiotherapy (30 x 20 Gy, or equivalent regimen, eg 33 x 18 Gy), with ≥ 90% of the planned radiation therapy dose delivered and concomitant TMZ chemotherapy (75 mg/m2), >66% of the planned doses administered.
7. Any toxicity attributable to recently completed chemoradiation must be resolved to the patient's baseline level or ≤ Grade 2 (except alopecia or lymphopenia).
8. Adequate bone marrow and organ function, defined by the following laboratory values: A. Absolute neutrophil count (ANC) ≥ 1000 cells/mm3 B. Platelet count ≥ 50,000 cells/mm3 C. Hemoglobin (Hgb) ≥ 8 g/dl D. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 x upper limit of normal (ULN) E. Total bilirubin ≤ 3 x ULN (unless gilbert's syndrome, then patients may be eligible if total serum bilirubin is ≤ 5.0 x ULN or direct bilirubin is ≤ 3 x ULN) F. Creatinine clearance (CrCl) as estimated by Cockcroft-Gault equation of ≥ 50 ml/min
9. Adequate coagulation function defined as PT (prothrombin time)/PTT (partial thromboplastin time) defined as either results within normal institutional values or not considered clinically significant <1.5 x ULN.
10. Non-pregnant, non-lactating females who are postmenopausal, surgically sterile (bilateral tubal ligation with surgery at least 6 weeks prior to study initiation or hysterectomy), or who agree to use effective contraceptive methods as defined by the protocol during the study and for 30 days after the last investigational treatment, see Appendix 1. Postmenopausal is defined as at least 12 months natural spontaneous amenorrhea and a serum follicle stimulating hormone (FSH) concentration ≥ 40 IU/L, or at least 6 weeks following surgical menopause (bilateral oophorectomy). See Appendix 1, females on HRT and whose menopausal status is in doubt will be required to use one of the non-estrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.
11. Women of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) pregnancy test within 7 days prior to first 5-ALA administration
12. Male patients must be surgically sterile (i.e., 3 months post- vasectomy) or willing to use a highly effective double-barrier contraception method (e.g., male condom with diaphragm or male condom with cervical cap) for the duration of the study and for at least 30 days following SDT treatment. Male patients must not donate sperm from the time of study drug dosing until 30 days following SDT treatment.
13. No anti-cancer treatment during adjuvant setting after completion of radiation therapy with anything other than temozolomide on Day 2 (+/-1 day) for 5 days per the approved Package Insert (PI).

Exclusion Criteria:

1. Any component of the tumor in the infratentorial location (cerebellar or brainstem tumors are excluded)
2. Bihemispheric disease or tumors that involve the bilateral corpus callosum, or disease burden involving the brain stem or cerebellum based on MRI post-gadolinium enhancement,
3. Multi- centric disease (enhancing or non-enhancing) or multi-focal disease (defined as 2 separate areas of contrast enhancement measuring at least 1 cm that are not contiguous and cannot be encompassed in sonication field on either fluid-attenuated inversion recovery (FLAIR) or T2 hyperintensity.
4. Leptomeningeal disease
5. 6. A diagnosis of glioscarcoma by histopathology Intent to undergo treatment with the tumor treating fields (TTF) at any time during the study, use prior to screening is permitted.

7. Corticosteroid use > 4 mg/day of dexamethasone (or equivalent), steroid dose should be stable or decreasing for ≥1 week prior to randomization 8. Inability to undergo MRI or receive gadolinium (Gd)-based contrast agents 9. Hypersensitivity to 5-ALA or porphyrins 10. Patient head size > 16.6 cm in breadth (max width of head, above the ears) and > 21.3 cm in length (front to back) to ensure fit within the helmet transducer array. 11. Skull voids/defects > 10 mm diameter if defect is open, or > 14 mm if defect is covered with titanium burr hole cover, titanium mesh, or similar repair hardware. Note, Longeviti Neuro Solutions or other sonolucent implants should be treated as open defects and therefore may not exceed 10 mm in diameter. 12. Hemorrhagic or ischemic stroke (including transient ischemic attacks) and central nervous system bleeding in the preceding 6 months that are not related to glioma surgery. History of prior intratumoral bleeding prior to screening is not an exclusion criterion; however, patients with a history of prior intratumoral or intracranial bleeding will undergo a non-contrast head CT to exclude acute bleeding. 13. Has any history of glioma, a concurrent malignancy, or malignancy within 3 years of randomization, unless definitive therapy is completed, with the exception of basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast that has completed curative therapy 14. Patients who have clinically significant cerebral edema requiring urgent intervention (e.g., surgery, initiation of steroids, escalating doses of steroids). 15. Patients with rapid clinical deterioration that, in the opinion of the investigator, is likely to worsen during the first cycle of treatment. 16. Any prior treatment for glioma, aside from surgical resection, and chemoradiation with TMZ. TTF is permitted prior to study entry. Agents used for diagnosis, imaging or visualization, even if investigational, are not exclusionary. Exclusionary treatments would include, but are not limited to: A. Stereotactic radiosurgery B. Placement of Gliadel® (carmustine; BCNU) wafers C. Any other intratumoral or intracavity treatment, D. Receipt of other chemotherapies, bevacizumab, immunotherapy (including vaccine) or investigational agents. 17. Acute or chronic types of porphyria. 18. Gastrointestinal disorder that negatively affects absorption. 19. Known active hepatitis B or C (Note: testing is not required). 20. Known human immunodeficiency virus (HIV) infection (Note: testing is not required). 21. Participation in another interventional clinical trial for GBM. (Observational studies are allowable) 22. Unable to avoid phototoxic drugs (e.g., St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulfonamides, quinolones, and tetracyclines) for 24 hours prior to and following 5- ALA administration. 23. Any other concurrent severe or uncontrolled concomitant medical condition that could compromise participation in the study (e.g., clinically significant pulmonary disease, cardiac disease, clinically significant psychiatric or neurological disorder, active or uncontrolled infection). 24. Women who are pregnant or breastfeeding 25. Patients with a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate and compare progression-free survival of patients by treatment arm | Up to 24 months

SECONDARY OUTCOMES:
Evaluate and compare overall survival of patients by treatment arm | Up to 24 months
  Key Secondary
Evaluate and compare survival at specific time points by treatment arm | 12, 18 and 24 months
Evaluate the number of participants with treatment-related adverse events as assessed by CTCAE by treatment arm | Up to 24 months
Evaluate time to next treatment for 5-ALA + LIDU SDT System | Up to 24 months

OTHER OUTCOMES:
Identify and evaluate prognostic and predictive factors (e.g. MGMT, extent of resection) for PFS | Up to 24 months
  Exploratory
Identify and evaluate prognostic and predictive factors (e.g. MGMT, extent of resection) for OS | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Albany Medical Center, Albany, New York
  - Northwell Health, Long Island City, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania